CLINICAL TRIAL: NCT05565014
Title: An Open Label, Randomized Controlled Clinical Study on the Safety and Efficacy of Virus Activated Killer Immune Cells (VAK) in the Treatment of Malignant Pleural and Peritoneal Effusion
Brief Title: Safety and Efficacy Study of Virus Activated Killer Immune Cells (VAK) for Malignant Pleural and Peritoneal Effusion
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheng Hu (Other)
Collaborators: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Sheng Hu, chief physician, Hubei Cancer Hospital
Organization: Hubei Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBCHC03
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Malignant Pleural Effusion; Malignant Peritoneal Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virus Activated Killer immune Cells（VAK） (Experimental): The VAK should be given once a week, three times a circle. The VAK could given 1 or 2 circle for each subject. The dosage of Pleural Effusion（more than 10^5/kg cells in 30-50mL solvent） differs from Peritoneal Effusion（more than 10^4/kg cells in 30-50mL solvent）
  Interventions: Drug: Virus Activated Killer immune Cells
- saline (Placebo Comparator): 50ml of saline was injected once a week,three times a circle.The saline could given 1 or 2 circle for each subject.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Virus Activated Killer immune Cells — The VAK made from Pleural Effusion should be given to treat Malignant Pleural Effusion.The VAK made from Peritoneal Effusion should be given to treat Malignant Peritoneal Effusion.
  Other Names: VAK
  Arms: Virus Activated Killer immune Cells（VAK）
Drug: Saline — The use of saline was the same as VAK group.
  Arms: saline

SUMMARY:
Theory of VAK：

1. Immune cells (T cells for example) of cancer subjects may be domesticated by the tumor microenvironment, and have low efficacy to kill cancer cells. They could be restimulated by virus antigen, and play a powerful tumor killing role while intrapleural to subjects.
2. Releasing of tumor-associated antigen could induce specific anti-tumor immune response.

Preparation of VAK：

1. Separate the immune cells and tumor cells from Malignant Pleural and Peritoneal Effusion.
2. Incubate the immune cells with inactivated viruses and tumor cells.
3. Wash to remove impurities.
4. Intrapleural the immune cells to patients

DETAILED DESCRIPTION:
There are a large number of immune cells in immune tolerance state in the tumor microenvironment. The theoretical basis of this clinical study is to use ultraviolet inactivated oncolytic herpes simplex virus type 2 (UV-oHSV2) to activate PBMC or immune cells in immune tolerance state in malignant pleural and peritoneal fluid in vitro, and to transfusion the activated immune cells back to the patient's peripheral blood or pleural and peritoneal fluid to kill tumor cells in malignant pleural and peritoneal fluid to further control the volume of malignant pleural and peritoneal fluid.

Our study indicated that UV-oHSV2 potently activated human peripheral blood mononuclear cells leading to increased antitumor activity in vitro and in vivo. We also found that UV-oHSV2 could induce NK cells (isolated from healthy donors' PBMC or patient pleural effusion) proliferation, secretion of IFN-γ. We further found that UV-oHSV2 could enhance NK cells (isolated from healthy PBMC or patient pleural effusion) antitumor ability in vitro and in vivo.

Based on the above research, we carried out an open, single center, prospective clinical trial to evaluate the safety and effectiveness of VAK cells in the treatment of malignant pleural and peritoneal effusions.

The detailed protocol as follow:

Isolation of lymphocytes from the patient's pleural effusions or ascites:

1. Add pleural fluid into a 50ml centrifuge tube, centrifuge at 400g, and discard the supernatant.
2. Resuspend the precipitate with 40ml of normal saline and pass through 70 μ M U.M and then rinse the cell filter once with 5ml physiological saline.
3. Discard the cell filter, and centrifuge the filtered cell suspension in the centrifuge tube at 400g for 5min. After centrifugation, discard the supernatant and resuspend the cell pellet with 5ml of normal saline.
4. Mix Ficoll upside down before use, take a new 15ml centrifuge tube and add 5ml Ficoll (suck with syringe).
5. Gently add 5-6ml cell suspension onto Ficoll layer.
6. Centrifuge 400g, 30-40min, 18 ℃ - 20 ℃, the centrifuge needs to be slowly raised and lowered, and the sudden stop braking setting should be closed.
7. Take the middle white membrane layer (lymphocytes) into a new centrifuge tube.
8. Add 3 times the volume of normal saline to the absorbed lymphocytes, resuspend the cells, centrifuge 400-500g, 10-15min, 18 ℃ - 20 ℃.
9. Repeat washing once, and the final precipitate is resuspended with 5ml serum-free medium (RPMI1640).
10. Take 20 μ L of cell suspension in EP tube, add equal volume of trypan blue staining solution, gently blow and count with cell counter.
11. In the process of planting the isolated immune cells, the cell culture density was controlled within the range of 106, and 10% autologous plasma was added.
12. Take 4ml of cell suspension for separate culture, and add the corresponding amount of inactivated virus to the remaining cell suspension with the infection number MOI = 1. The calculation formula is as follows: volume of uv-oh2 added = (1 × Number of cells added per well plate or bottle / oh2 virus titer)
13. After the immune cells are planted, they are placed in a 5% CO2 incubator for 36h-48h.

After cell culture, 30-50ML of prepared lymphocytes (qualified by PCR sterility test and endotoxin test) were infused into the chest and abdominal cavity of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign informed consent;
2. Pathological confirmed advanced malignant tumor with malignant pleural or peritoneal effusion;
3. Vital signs stable, Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2;
4. Age ≥ 18 years old, gender unlimited;
5. Expected survival period more than 3 months;
6. Subjects agree to take effective contraceptive measures at the time of enrollment and within 4 months after enrollment. The pregnancy test of female patients must be negative;
7. Sufficient bone marrow, liver and kidney functions. Laboratory tests within 7 days before the first drug use meet the following requirements:

   * Coagulation function: APTT ≤ 1.5 × ULN, while INR or PT ≤ 1.5 × ULN (not receiving anticoagulant therapy); ② Blood routine examination: Hgb ≥ 80g / L, WBC > 3 × 10^9/L、NEU≥1.0 × 10^9/L、PLT≥80 × 10^9/L;
   * Liver function: total bilirubin ≤ 1.5 times the upper limit of normal value (ULN); AST and alt ≤ 2.5 times ULN (if abnormal liver function is mainly caused by tumor infiltration, it can be ≤ 5 times ULN; alkaline phosphatase ≤ 2.5 times ULN; ④ Renal function: bun and Cr ≤ 1.5 times ULN, creatinine clearance ≥ 40ml / min (calculated by Cockcroft Gault formula).

Exclusion Criteria:

1. Subjects requiring emergency treatment due to intestinal obstruction or vascular compression;
2. Subjects with active hemolytic anemia;
3. Subjects with active central nervous system metastases were excluded, except those with brain metastases or asymptomatic cancer cells found in cerebrospinal fluid;
4. Pregnant or lactating female;
5. Systemic active infection, serious coagulation disorder or serious heart, respiratory and immune system diseases;
6. Congenital or acquired immune function defects (such as HIV infection), hepatitis B infection (HBV-DNA ≥ 10 ^ 4 / ml), hepatitis C infection (HCV antibody and HCV RNA positive);
7. Subjects who had serious infection within 4 weeks before the first medication were excluded, including but not limited to infectious complications, bacteremia and severe pneumonia requiring hospitalization;
8. Subjects with active autoimmune diseases or a history of autoimmune diseases that may recur, but the following are not excluded:

   * Type 1 diabetes
   * Hypothyroidism (if controlled by hormone replacement therapy only)
   * Controlled celiac disease ④ Skin diseases without systemic treatment (such as vitiligo, psoriasis, alopecia) ⑤ Any other disease that does not recur without external triggers.
9. Those who had severe hypersensitivity to the drugs used in this protocol in the past;
10. Subjects who are ready for or have previously received tissue / organ transplantation;
11. Subjects with large pericardial effusion were excluded;
12. Exclude those who have suffered from other malignant tumors within 2 years, except for cervical carcinoma in situ, low-risk gastrointestinal stromal tumor, skin basal cell carcinoma, skin squamous cell carcinoma, thyroid papillary carcinoma and breast ductal carcinoma in situ that have been effectively removed;
13. Exclude subjects who have been vaccinated or will be vaccinated with live vaccine within 4 weeks before the first administration;
14. Other circumstances that the investigator considers inappropriate for clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs | 28 days after the last treatment.
  Incidence of adverse events (AEs) and serious adverse events (SAEs) graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
ORR of Malignant Pleural and Peritoneal Effusion by WHO 1997 | 28 days after the last treatment.
  The volume of pleural and peritoneal effusion was measured by volume software of spiral CT machine to determine the change of pleural and peritoneal effusion volume before and after treatment. ORR=PR+CR.
Progression Free Survival | up to 1 year.
  Progression free survival from day 1 of treatment until death or progression.
Overall Survival | up to 2 year.
  Overall survival from day 1 of treatment until death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No